CLINICAL TRIAL: NCT07256626
Title: Tune Up Your Back: Soundwave Wellness Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Efforia, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 37378
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-11

CONDITIONS: Pain, Back
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Intervention Model Description: Single Arm observational where participants act as their own control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single arm where participants act as their own control (Experimental): Single arm where participants act as their own control
  Interventions: Device: WAVWatch 2.0

INTERVENTIONS:
Device: WAVWatch 2.0 — The WAVwatch sound frequency therapy device employs acoustic waves absorbed through the skin to promote wellness, with manufacturers and users reporting minimal safety risks

SUMMARY:
Looking to support your back mobility and overall comfort? Join our study exploring WAVwatch 2.0, an innovative soundwave therapy device. This non-invasive technology is designed for individuals who want to maintain easy movement and flexibility without constantly reaching for over-the-counter options. By joining, you'll discover how this gentle approach may help support everyday back comfort, mobility, and flexibility.

DETAILED DESCRIPTION:
This remotely administered decentralized trial is designed to methodically explore the efficacy of WAVwatch 2.0, a non-invasive device that leverages soundwave therapy, in enhancing back comfort and flexibility. In the wake of increasing reliance on temporary solutions for back tension and stiffness, this study emerges as a pivotal investigation into whether soundwave therapy can offer a sustainable pathway to maintaining ease of back movement and overall wellness.

The primary objective of this online trial is to facilitate participants in understanding the potential benefits of WAVwatch 2.0 on their daily comfort, range of motion, and general quality of life. Through this exploratory journey, participants will receive personalized insights, enabling a comprehensive understanding of how soundwave therapy might influence their back comfort and mobility. This initiative aims not only to assess the device's ability to support back wellness but also to empower participants with knowledge about alternative, non-invasive options for enhancing their quality of life.

Focusing on the experiential changes in ease of movement, daily activities, and overall wellness, the study intends to rigorously evaluate and document the impact of WAVwatch 2.0 on participants. By doing so, it seeks to offer a detailed perspective on the device's effectiveness in promoting back health and comfort. The trial is committed to providing participants with a clear, personalized overview of how soundwave therapy could integrate into their wellness routines, potentially redefining approaches to back care.

The significance of this remotely conducted trial extends beyond individual benefits, aiming to contribute to the broader understanding of non-invasive back care solutions. By examining the outcomes of using WAVwatch 2.0 for back comfort and mobility, the study aspires to challenge and expand current perspectives on managing back tension and stiffness, offering new insights into the role of soundwave therapy in daily wellness practices.

It is important to note that throughout this trial, the PROMISE and ROMISE scales will serve as key tools in assessing participants' quality of life, comfort, and ease of movement. These scales, while integral to evaluating the benefits of WAVwatch 2.0, are not utilized as diagnostic instruments but as means to gauge the subjective experience of participants, thereby enriching the study's findings on the feasibility of soundwave therapy as a supportive measure for back wellness.

ELIGIBILITY:
Inclusion Criteria:

* Can read and understand English.
* US resident.
* Willing and able to follow the requirements of the protocol.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
PROMIS® Item Bank/Scale v.2.0 - Pain Behavior Survey | Change from baseline (Day 1-3) in pain behavior at 4 weeks after the start of the intervention (Day 27-33)
  This survey aims to understand individual behaviors and reactions when experiencing pain within the past 7 days.
Quality of Life and Health Survey | Change from baseline (Day 1-3) in quality of life at 4 weeks after the start of the intervention (Day 27-33)
  This survey asks about your feelings towards your quality of life, health, and various areas of your life. It covers your experiences and feelings in the past four weeks. Please choose the answer that appears most appropriate.
ROMIS® Numeric Rating Scale v.1.0 - Pain Intensity 1a | Change from baseline (Day 1-3) in pain intensity at 1 week after the start of the intervention (Day 4-10)
  This survey is designed to understand the level of pain experienced by the participant in the past 7 days. The responses will help in assessing the pain intensity from no pain to worst imaginable pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Efforia, New York, New York, United States

REFERENCES:
- See also: Additional information and join instructions on Efforia — https://app.efforia.com/wp-admin/admin.php?page=llms-course-builder&course_id=37378